CLINICAL TRIAL: NCT07060677
Title: Effectiveness of Immersive Virtual Reality Combined With Occupational Therapy in Reducing Fall Risk and Frailty Among Older Adults
Acronym: VIRTO-FRAIL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Cristina García-Bravo, Principal Investigator, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 080520254252025
Record Dates: First submitted 2025-06-19; First posted 2025-07-11 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Frailty Syndrome; Older Adults, Balance; Fall Prevention in Healthy Aging
Keywords: Inmersive Virtual Reality; Occupational Therapy; Frailty Sindrome; Fall Prevention; Older Adults; Pre-Frailty; Quality of Life
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: Control Group (CG), which received their usual sessions of conventional occupational therapy, and an Experimental Group (EG), which received therapy with Inmersive Virtual Reality, plus their conventional occupational therapy sessions.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (EG) (Experimental): Experimental Group (EG), which received therapy with Inmersive Virtual Reality, plus their conventional occupational therapy sessions.
  Interventions: Procedure: Inmersive Virtual Reality; Procedure: Conventional occupational therapy sessions
- Control Group (CG) (Active Comparator): Control Group (CG), which received their usual sessions of conventional occupational therapy.
  Interventions: Procedure: Conventional occupational therapy sessions

INTERVENTIONS:
Procedure: Inmersive Virtual Reality — Participants will receive a intervention of immersive virtual reality using Meta Quest 3 and the Kinesix XR platform. Sessions will take place twice per week for 8 weeks. The IVR component will focus on balance and mobility through interactive, immersive environments designed to enhance engagement, adherence, and functional outcomes. This multimodal approach aims to reduce fall risk and frailty while improving motivation and quality of life in older adults.
  Arms: Experimental Group (EG)
Procedure: Conventional occupational therapy sessions — Participants will receive conventional occupational therapy only, with sessions conducted twice per week for 8 weeks. The intervention will focus on cognitive stimulation, manipulative skill training, and psychomotor exercises, all adapted to the functional level of each participant. Activities aim to maintain or improve autonomy, balance, and coordination, following established occupational therapy guidelines for older adults. No immersive virtual reality or digital technology will be included in this group. This control condition allows for comparison with the experimental group to evaluate the added value of immersive virtual reality in fall risk and frailty reduction.

SUMMARY:
Population aging is a growing global phenomenon that poses significant challenges to healthcare systems, particularly in preventing falls and managing frailty among older adults. Falls remain a leading cause of morbidity and mortality in this population, affecting approximately one-third of individuals over 65 each year. At the same time, frailty syndrome (FS)-a clinical condition marked by progressive decline in physical and cognitive function-significantly increases the risk of falls, disability, and dependency. Pre-frailty, an intermediate and reversible stage, offers a key opportunity for preventive interventions.

Scientific evidence supports the effectiveness of interdisciplinary approaches to address frailty and fall prevention. In this context, occupational therapy plays a central role by promoting functional autonomy through meaningful activities. However, traditional approaches may be limited in individuals with low motivation or mild cognitive impairment. Therefore, integrating innovative technologies such as immersive virtual reality (IVR) emerges as a promising therapeutic strategy.

IVR enables users to interact with simulated three-dimensional environments, enhancing cognitive stimulation, motor training, and treatment adherence. Modern devices like the Meta Quest 3 headsets provide accessible, safe, and adaptable immersive experiences, with reported benefits in balance, gait, attention, and motivation. Nonetheless, no studies to date have specifically evaluated the effectiveness of this technology when combined with conventional occupational therapy to reduce fall risk and frailty in older adults.

This project proposes a pilot randomized controlled trial (RCT), lasting 5 months, using a single-blind, parallel-group design. It will be conducted at the Bouco Madrid Ferraz Residential Center (Madrid, Spain), following CONSORT 2010 methodological guidelines. The primary aim is to assess the efficacy of a combined intervention using IVR through Meta Quest 3 headsets and occupational therapy, compared to conventional occupational therapy alone, in reducing fall risk, improving frailty status, enhancing quality of life, and increasing rehabilitation motivation in older adults.

The sample will include 30 participants (15 per group), selected based on specific inclusion and exclusion criteria. Participants will be randomly assigned to a control group (CG), receiving standard occupational therapy, or to an experimental group (EG), receiving a combined intervention of occupational therapy and IVR using the Kinesix XR platform, which is designed to enhance balance.

The intervention will last 8 weeks, with two one-hour sessions per week. The experimental group will receive 30 minutes of occupational therapy and 30 minutes of IVR per session. Assessments will be conducted at baseline, post-intervention, and at a 3-month follow-up using validated scales to measure fall risk, balance, frailty level, quality of life, and satisfaction.

Data will be pseudonymized, statistically analyzed using SPSS, and managed in compliance with the European General Data Protection Regulation (EU 2016/679). The small sample size reflects the exploratory nature of the study, aimed at assessing feasibility, safety, and preliminary outcomes prior to conducting a larger-scale trial.

Ultimately, this project aims to provide initial evidence on an innovative intervention for older adults by integrating digital tools with conventional therapeutic approaches. If proven effective, the VIRTO-FRAIL model could lay the groundwork for new strategies in geriatric rehabilitation and fall prevention.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 years or older
* Regularly attending rehabilitation treatment at the Bouco Madrid Ferraz Residence
* Having the ability to walk with or without assistive devices
* Presenting sufficient cognitive capacity to understand instructions (score ≥ 24 on the MMSE)
* Agreeing to participate voluntarily
* Signing the informed consent form.

Exclusion Criteria:

* Having a diagnosis of a severe neurological disease (such as advanced Parkinson's disease or ALS, among others)
* Having a history of epilepsy or seizures (due to potential adverse effects with VR)
* Experiencing cardiovascular instability or having a medical contraindication for physical activity
* Presenting vestibular disorders
* Participating in other similar intervention programs during the same period
* Being unable to use virtual reality glasses due to intolerance or dizziness
* Not agreeing to participate voluntarily in the study and/or not signing the informed consent form.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2025-09-25 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Functional Independence Measure (FIM) | Pre-intervention, post-intervention (up to 1 week) and follow-up (3-month)
  An instrument that assesses the level of functional independence in activities of daily living. It provides information primarily on motor and cognitive performance through 18 items. Each item is scored from 1 to 7, with higher scores indicating greater functional independence. The assessment is conducted through task observation and interview.
Functional Reach Test | Pre-intervention, post-intervention (up to 1 week) and follow-up (3 month)
  This test measures the maximum distance an individual can shift their center of gravity towards the limits of their base of support. In a relaxed standing posture, with feet hip-width apart, the participant is asked to flex the shoulder to 90 degrees and keep the hand extended. They must then reach forward as far as possible. The examiner records the furthest distance the center of gravity is displaced. Two practice trials and three recorded trials are conducted, with the average of the three being the final score. The result is recorded in centimeters.
Timed 'Up and Go' (TUG) | Pre-intervention, post-intervention (up to 1 week) and follow-up (3-month)
  This test measures the time it takes a person to rise from a chair, walk 3 meters, turn around, return to the chair, and sit down again. It evaluates balance and gait speed. The score is recorded in seconds.
Clinical Frailty Scale (CFS) | Pre-intervention, post-intervention (up to 1 week) and follow-up (3-month)
  A clinical tool used to assess the level of frailty in older adults. It is based on a 9-point scale, where patients are classified from 1 (very fit) to 9 (terminally ill), reflecting increasing severity of frailty. Higher scores indicate worse outcomes, representing greater vulnerability and dependency. The evaluation incorporates physical and cognitive function, as well as the level of dependency, to estimate a patient's vulnerability to stressors.
Kinesix Virtual Reality Therapeutics© Functional Assessment Scale | Pre-intervention, post-intervention (up to 1 week) and follow-up (3-month)
  Designed to objectively measure and analyze a person's performance in specific tasks. This tool evaluates upper limb reach, balance, and other key functional capacities, providing valuable information for establishing a starting point and tracking patient progress over time.
  Scores on the Kinesix VR Therapeutics© Functional Assessment Scale range from 0 to 100, with higher scores indicating better functional performance and a more favorable outcome. A score of 0 reflects minimal or no functional ability, while a score of 100 indicates optimal or fully restored function.
  This scale is intended for use by trained clinicians and therapists to monitor patient progress over time, assess the effectiveness of VR interventions, and support individualized treatment planning.
World Health Organization Quality of Life - BREF (WHOQOL-BREF) | Pre-intervention, post-intervention (up to 1 week) and follow-up (3-month)
  A self-administered questionnaire that evaluates overall perception of quality of life and general health status. It consists of four domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF consists of 26 items that measure four domains: Physical Health, Psychological Health, Social Relationships, and Environment. Each item is rated on a 5-point Likert scale, and domain scores are transformed to range from 0 to 100, in accordance with WHO scoring guidelines.
  Higher scores on the WHOQOL-BREF indicate a better quality of life. A score of 0 represents the lowest possible quality of life in a domain, while a score of 100 reflects the highest possible perceived quality of life.
  The WHOQOL-BREF provides a comprehensive yet efficient assessment of well-being and is validated across a wide range of cultures and populations.

SECONDARY OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | Post-intervention (up to 1 week)
  A self-administered questionnaire consisting of 8 items that assess satisfaction with the care and quality of services received, as well as how well the intervention met the patient's expectations. Responses are scored from 1 to 4, with a maximum score of 32; higher scores indicate greater satisfaction. The Spanish adaptation of the questionnaire has shown adequate psychometric properties and preserves the characteristics of the original version, making it suitable for assessing satisfaction with healthcare services in the Spanish population. The CSQ-8 will be administered to both treatment groups in this study.
System Usability Scale (SUS) | Post-intervention (up to 1 week)
  A usability evaluation scale used to assess the effectiveness of virtual reality in healthcare settings. It includes 10 items that cover various aspects of the user's experience with the technology, such as ease of use, efficiency, and overall satisfaction. Responses range from "strongly agree" to "strongly disagree."

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Universidad Rey Juan Carlos, Alcorcón, Marid
  - Residencia Bouco Madrid Ferraz, Madrid

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/77/NCT07060677/ICF_000.pdf